CLINICAL TRIAL: NCT04195165
Title: The Effect of Sitting and Moderate Exercise on Plasma Insulin and Glucose Responses to an Oral Glucose Tolerance Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael B. Dial, Graduate Student, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-08-0011
Record Dates: First submitted 2019-09-24; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Sedentary Behavior; Insulin Sensitivity; Sedentary Lifestyle
Keywords: glucose tolerance; exercise; insulin sensitivity
MeSH Terms: conditions — Sedentary Behavior; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIT (Experimental): Subject will be asked to take <3,000 steps for two intervention days prior to an oral glucose tolerance test on the third day.
  Interventions: Behavioral: SIT
- SIT+EX (Experimental): Subject will be asked to take <3,000 steps for two intervention days. On the evening of the second intervention day, the subject will cycle for one hour at 65% of VO2peak. The subject will undergo an oral glucose tolerance test on the morning of the third day.
  Interventions: Behavioral: SIT; Behavioral: EX
- ACTIVE+EX (Experimental): Subject will be asked to take >10,000 steps for two intervention days. On the evening of the second intervention day, the subject will cycle for one hour at 65% of VO2peak. The subject will undergo an oral glucose tolerance test on the morning of the third day.
  Interventions: Behavioral: ACTIVE; Behavioral: EX

INTERVENTIONS:
Behavioral: SIT — For the SIT and SIT+EX conditions, the subject will be asked to take <3,000 steps. This is meant to achieve ~12-13 hours of sitting per day, are the investigators are measuring the effect of inactivity and exercise on insulin sensitivity.
  Arms: SIT; SIT+EX
Behavioral: ACTIVE — For the ACTIVE+EX condition, the subject will be asked to take >10,000 steps for the two intervention days. This is meant to simulate an active lifestyle.
  Arms: ACTIVE+EX
Behavioral: EX — The SIT+EX and ACTIVE+EX conditions will include an exercise bout on the evening of the second intervention day, and have the oral glucose tolerance test the next morning.
  Other Names: Exercise
  Arms: ACTIVE+EX; SIT+EX

SUMMARY:
The investigators hypothesize that cycling for 1 hour of exercise at 65% peak oxygen consumption (VO2peak) after sitting >13 hr/day (SIT+EX) will not be different in postprandial plasma insulin responses compared to the control of only sitting (SIT). Furthermore, the investigators hypothesize that the SIT and SIT+EX groups will have a less favorble insulin response compared to the physically active group after performing the same 1-hour exercise bout (ACTIVE+EX).

DETAILED DESCRIPTION:
Twelve healthy, untrained male and female participants will complete three different trials in a randomized, crossover design, each occurring over 4 days with a 3-4 day interval between the trials. Each trial consists of 3 phases. The first two days will serve as a control phase (C1) that will allow for familiarization, followed by a 2-day intervention phase consisting of 2 days of sitting 13 h/d for both groups (D1- D2) (SIT+EX and ACTIVE+EX). On the evening of Day 2 the SIT+EX and ACTIVE+EX groups will cycle for 1 hour at 65% of VO2peak. On the morning of Day 3 participants in all conditions will ingest a drink containing 75-g of glucose and undergo a two-hour oral glucose tolerance test (OGTT). For all trials, participants will refrain from any exercise other than that described for the study.

One week prior to the initiation of the first trial, participants will visit the Human Performance Laboratory (HPL) for a 10 min exercise test to measure peak oxygen uptake while cycling (VO2peak). On the same day, participants will be instrumented with an activity monitor worn on their thigh to record time sitting, standing and lying as well as step count (activPal). During the two control day (C1), participants will be asked to refrain from any planned exercise but will be asked to walk or move between 6,000 - 7,500 steps per day, which is considered to be 'low level of physical activity'(31). During the intervention days (D1-D2), those completing SIT and SIT+EX conditions will be asked to remain seated throughout much of the day and achieve <3,000 steps, while those completing the ACTIVE+EX condition will be asked to break up their sitting with low-intensity physical activity, not exercise, and achieve >10,000 steps. However, the only difference between trials is that at 18:00 h during SIT+EX and ACTIVE+EX they will cycle for 1-hr at 65% VO2peak.

On the day of the OGTT (D3), participants will report to the laboratory at 07:00 h. Body weight will be measured. They will lay down for 5 minutes and a catheter will be inserted into an antecubital vein and a fasting blood sample will then be collected 10 min before consumption of high-glucose drink (75 g) composed of water and glucose monohydrate. Approximately 5 ml of blood will be collected at 10, 20, 30, 60, 90 and 120 min after ingestion. Approximately 60 ml of blood will be sampled during each of the three trials and thus the total will amount to approximately 180 ml (6 ounces, 12 tablespoons). This amounts to approximately 2-4% of a person's total blood volume.

All blood samples collected will be transferred to K2 EDTA collection tubes, centrifuged at 2,000 g for 15 minutes at 4◦C and then stored in -80◦C freezer until later analysis. During OGTT, participants will sit quietly reading, watching movies, and/or surfing the Internet. Participants will also be asked to keep a consistent sleep/wake cycle during the trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, untrained/recreationally active men and women.
* Women must not be pregnant or post-menopausal.

Exclusion Criteria:

* Heart problems or coronary artery disease
* Hypertension
* Lung or respiratory problems
* Chest pain, fainting, or heart palpitations during exercise, or told to give up sports because of health problems.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-23 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Up to 4 weeks after data completion
  The investigators will measure glucose and insulin levels from data collected during the oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Dial, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No